CLINICAL TRIAL: NCT05758441
Title: Mentoring to be Active: Peer Mentoring to Mitigate Obesity and Extreme Obesity in Rural Appalachian Children
Brief Title: Mentoring to be Active for Rural Appalachia Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GR130196; 11-22-ICTSN-30 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2023-02-16; First posted 2023-03-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Physical Activity; Exercise; Body Composition
Keywords: Physical Activity, Body Composition, Health Behavior
MeSH Terms: conditions — Motor Activity; Health Behavior

STUDY DESIGN:
Intervention Model Description: For this community-based study, a stratified randomized-controlled clinical trial will evaluate MPBA+F among 7/8th grade children with overweight or obesity recruited during years 1 and 2 of the study from rural Appalachian counties. Stratification by biological sex to have equal numbers of males and females will occur. Investigators will recruit 288 children to participate. Half will be randomized to receive MPBA+F; the other half will receive a comparison program of 10 weekly, self-guided modules from mailed to their home. By following participants from the start of 7th grade (baseline) through the middle of 8th grade, longer-term effects on PA outcomes and body composition can be determined. Differences in outcomes are explored by examining sub-group differences on effects. A sub-set of parents from both study conditions will be recruited (72 parents from each condition) to provide child assessments of perceived PA behaviors and perceived child health.
Who Masked: Outcomes Assessor
Masking Description: Trained research assistants who will collect data and survey measures are blinded to study condition of each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mentoring to be Active plus Family (MPBA+F) (Experimental): For the first phase, ten peer-mentoring sessions (1 day/week for 45 minutes each week) delivered virtually with a Project Leader, five peer mentors, and 8-10 mentees with 1:2 mentor/mentee ratios. Each session consists of a 10-15 minute content lesson followed by 20-30 minutes of guided practice, social support, feedback, and personal goal-setting for the following week in small peer mentor/mentee "break-out" rooms. Mentees track activities and efforts towards meeting personal goals. Parents return their child's weekly completed 'Tracker" forms either electronically via the secure, password-protected project website or (if they prefer) by regular pre-paid mail service. The reinforcement component of MPBA+F is a guided, parent-directed 6-module (0nce a month for 6 months) program for parents/guardians to further support the child's home-based PA. Child participants assigned to MPBA will be provided the modules.
  Interventions: Behavioral: Mentoring to be Active plus Family
- Tracking Health and Fitness (Active Comparator): Half of child participants will receive "Tracking your Health and Fitness", a comparison program of 10 weekly, self-guided modules from Ohio State University (OSU) Extension mailed to their home.
  Child participants assigned to the "Tracking Health and Fitness" program (comparison group) may voluntarily participate in a 6-month rewards-based self-regulation program to encourage sustainability of weekly PA.
  Interventions: Behavioral: Tracking Health and Fitness

INTERVENTIONS:
Behavioral: Mentoring to be Active plus Family — Ten, structured peer mentoring sessions (once a week) covering new content each week and guided skill-building and practice. The MPBA sessions target increasing daily physical activity and replacing sugary drinks with water for hydration. Mentoring sessions are conducted virtually. A 6-month family reinforcement program follows with a reinforcement packet sent to child participants' homes once a month.
  Other Names: MPBA
  Arms: Mentoring to be Active plus Family (MPBA+F)
Behavioral: Tracking Health and Fitness — 10 self-guided, self-paced modules mailed to child participants home.
  Arms: Tracking Health and Fitness

SUMMARY:
The innovative MPBA+F begins with peer-to-peer mentoring followed by structured parental/family support for long-term reinforcement of PA behaviors. Building and reinforcing skills, MPBA+F mitigates resource stressors and strengthens protective factors by providing culturally appropriate knowledge and skills to improve the sustainability of physical activity at home without the use of exercise equipment. By strengthening social support through peer and friendship networks and family-based support, MPBA+F responds to the unique needs of rural Appalachians in a culturally responsive way. This study targets physical activity among children with overweight, obesity, or extreme obesity because rural Appalachian communities identify sedentary activity as a key contributor to the high rates of obesity and diabetes risk among youth.

DETAILED DESCRIPTION:
Appalachians die more frequently and at younger ages from obesity-related conditions than those living elsewhere. High prevalence of overweight, obesity, and extreme obesity in Appalachian children increases the severity of diabetes. In rural Appalachia, the diabetes mortality rate is 11% higher than the national rate.Over the course of two years, this study will test the effects of the Mentored Planning to be Active + Family intervention on physical activity outcomes (MVPA, exercise "bouts", sedentary behavior) and health outcomes (body composition: BMI, body fat, % body fat, weight) among rural Appalachian 7/8th grade children suffering from overweight and obesity. Having teens deliver the content via structured peer mentoring increases social support, motivation, and self-regulation to sustain PA behaviors to improve health outcomes as children enter high school. Using local residents for intervention delivery leverages rural Appalachians' preference to receive health information via established social networks and extends delivery of the program into the community. This study is a community-based randomized controlled trial targeting 7th grade students in rural Appalachia. Half (n = 144) will receive MPBA+F; the other half (n = 144) will receive self-guided (usual care) modules. Tenth-grade (n = 73) students from the same rural Appalachian counties will serve as peer mentors delivering MPBA for the peer mentoring group. Parents will provide a family reinforcement program during 8th grade and provide assessments of child behaviors and health outcomes. The long-term goal is to reduce the high rates of OW, OB/EO and type 2 diabetes in Appalachia youth through effective, sustainable interventions. Improving self-regulation, self-efficacy, and social support to increase intentional exercise and MVPA among underserved youth suffering from early-onset OB/EO builds healthier lifestyle behaviors at a critical development time.

ELIGIBILITY:
Inclusion Criteria:

Children:

* enrolled in 7th grade at the start of the study,
* have a body mass index percentile of 85th or greater for age and gender,
* not under medical care for OB or type 1 diabetes,
* have reliable internet connection at home,
* have access to a computer, laptop or tablet at home,
* not expected to move from the participating county before the conclusion of the study.

Parents:

* read at a 5th grade-level,
* speak English,
* have a home-mailing address (not PO box),
* have a working telephone number, and
* are not expected to move from the participating county before study conclusion.

High school peer mentors:

* are in either 10th or 11th grade at the start of the recruitment,
* reside in a targeted county,
* interested in working with peers, supporting others, and striving to cultivate their own health-supportive behaviors,
* have reliable internet connection at home,
* have access to a computer, laptop or tablet at home,
* are not expected to move before the intervention ends,
* can speak English,
* are recommended by a teacher, school advisor, or counselor.

Exclusion Criteria:

Child:

* not in 7th grade at the start of the study.
* not able to read or Speak English;
* not classified as either overweight or obese at start of study.

Parents :

- not able to read or speak English.

High school peer mentors:

- cannot speak and read English.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2026-11-14 (Estimated); Study Completion 2026-11-14 (Estimated)

PRIMARY OUTCOMES:
Change in Daily Physical Activity | 7 days- collected at baseline, at week 12 when mentoring sessions end, and at 9 months when the reinforcement program ends
  Daily levels of moderate and vigorous physical activity collected by accelerometry.

SECONDARY OUTCOMES:
Change in Body Composition | baseline, at 12 weeks when mentoring sessions end, and at 9 months when the reinforcement program ends.
  Anthropometric (body composition- raw weight, BMI, body fat) using the Tanita 430-DCU Body Composition Analyzer

OTHER OUTCOMES:
Change in Parent Perceptions of Child's Physical Activity Behaviors | Baseline and at 9 months when the reinforcement program ends.
  8-item PROMIS instrument measures the parent's perceptions of their child's performance of physical activity over the past 7 days. Physical actions reflect the levels of bodily movement ranging from simple static behaviors with minimal muscle activity to more complex activities requiring dynamic or sustained muscle activity and greater movement of the body.
Change in Parent Perceptions of Child's General Health | Baseline and at 9 months when the reinforcement program ends.
  7-item PROMIS Global Health instrument measures parent perceptions of their child's overall general health, physical health, mental health, social health and quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University College of Nursing, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
The American Diabetes Association policies and guidance for availability and sharing of research results and resources will be followed. All data that can be shared without compromising human subject protections will be shared to an approved open data repository as required. Study-related data will be anonymized, catalogued, and stored per federal guidelines and university policies. A public use, de-identified dataset will be available to qualified investigators upon request after analyses have been conducted and findings have been published. All identifiers will be removed. A request in writing, stating intended use must be submitted. Data sets will be accompanied by a data dictionary, both derived and raw data. The most cost-effective means for sharing data will be followed after a data sharing agreement has been reached. Curricular materials will be provided at no charge.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 6 months of publication or 18 months if results are not published.
Access Criteria: A written request for any study data, protocols or other materials must be sent to Principal Investigator. Once approved, materials will be made available by agreement.

REFERENCES:
- [Derived] Smith LH, Petosa RL, Tan A, Shankle S, Phosri Y. Randomised trial of Mentored 'Planning to be Active+Family' [MPBA+F] for Appalachian youth at risk for diabetes: virtual delivery protocol. BMJ Public Health. 2024 Nov 2;2(2):e000798. doi: 10.1136/bmjph-2023-000798. eCollection 2024 Dec. PMID 40018636